CLINICAL TRIAL: NCT05806320
Title: The Effect of Simulated Intrauterine Sound Applied to Preterms on Heart Rate, Oxygen Saturation and Comfort Level
Brief Title: The Effect of Simulated Intrauterine Sound Applied to Preterms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Birsen Mutlu, Associate Professor, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IUC-B-M-001
Record Dates: First submitted 2023-03-02; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Neonatal Intensive Care; Preterm
Keywords: Sound
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intrauterine Sound Listening Group 1 (Experimental): This group consisted of 15 infants with 26-32,6 GW. A total of one hour of noise measurement was made inside and outside the incubator before, during and after the procedure. The babies were listened to the sound obtained in 3 time periods. If the baby is fed enterally, the feeding of the baby was completed at 10.15/13.00/16.15 before the application, the baby was placed in the prone position and the baby was rested for 30 minutes to ensure gastric emptying. Before the procedure, the baby was watched with a monitor device and recorded on video between 10.45-11.00/13.30-13.45/16.45-17.00. During the baby procedure, uterine sound was listened to the baby in the prone position monitored with a monitor device and recorded on video between 11:00-11.30/13.45-14.15/17.00-17.30 hours. After the procedure, the baby was watched with a monitor device and recorded on video between 11.30-11.45/14.15 and 14.30/17.30-17.45.
  Interventions: Other: Intrauterine Sound Listening Group 1
- Intrauterine Sound Listening Group 2 (Experimental): This group consisted of 15 infants with 33-36,6 GW. A total of one hour of noise measurement was made inside and outside the incubator before, during and after the procedure. The babies were listened to the sound obtained in 3 time periods. If the baby is fed enterally, the feeding of the baby was completed at 10.15/13.00/16.15 before the application, the baby was placed in the prone position and the baby was rested for 30 minutes to ensure gastric emptying. Before the procedure, the baby was watched with a monitor device and recorded on video between 10.45-11.00/13.30-13.45/16.45-17.00. During the baby procedure, uterine sound was listened to the baby in the prone position monitored with a monitor device and recorded on video between 11:00-11.30/13.45-14.15/17.00-17.30 hours. After the procedure, the baby was watched with a monitor device and recorded on video between 11.30-11.45/14.15 and 14.30/17.30-17.45.
  Interventions: Other: Intrauterine Sound Listening Group 2
- Control Group 1 (No Intervention): This group consisted of 15 infants with 26-32,6 GW. A total of one hour of noise measurement was made inside and outside the incubator before, during and after the procedure. Babies in this group were followed up at specified time intervals without any intervention.
  If the baby is fed enterally, the feeding of the baby was completed at 10.15/13.00/16.15 before the application, the baby was placed in the prone position and the baby was rested for 30 minutes to ensure gastric emptying. The baby was watched with a monitor device and recorded on video between 10.45-11.00/13.30-13.45/16.45-17.00 hours; 11:00-11.30/13.45-14.15/17.00-17.30 hours; 11.30-11.45/14.15- 14.30/17.30-17.45.
- Control Group 2 (No Intervention): This group consisted of 15 infants with 33-36,6 GW. A total of one hour of noise measurement was made inside and outside the incubator before, during and after the procedure. Babies in this group were followed up at specified time intervals without any intervention.
  If the baby is fed enterally, the feeding of the baby was completed at 10.15/13.00/16.15 before the application, the baby was placed in the prone position and the baby was rested for 30 minutes to ensure gastric emptying. The baby was watched with a monitor device and recorded on video between 10.45-11.00/13.30-13.45/16.45-17.00 hours; 11:00-11.30/13.45-14.15/17.00-17.30 hours; 11.30-11.45/14.15- 14.30/17.30-17.45.

INTERVENTIONS:
Other: Intrauterine Sound Listening Group 1 — This group consisted of 15 infants with 26-32,6 GW. A total of one hour of noise measurement was made inside and outside the incubator before, during and after the procedure. The babies were listened to the sound obtained in 3 time periods. If the baby is fed enterally, the feeding of the baby was completed at 10.15/13.00/16.15 before the application, the baby was placed in the prone position and the baby was rested for 30 minutes to ensure gastric emptying. Before the procedure, the baby was watched with a monitor device and recorded on video between 10.45-11.00/13.30-13.45/16.45-17.00. During the baby procedure, uterine sound was listened to the baby in the prone position monitored with a monitor device and recorded on video between 11:00-11.30/13.45-14.15/17.00-17.30 hours. After the procedure, the baby was watched with a monitor device and recorded on video between 11.30-11.45/14.15 and 14.30/17.30-17.45.
  Arms: Intrauterine Sound Listening Group 1
Other: Intrauterine Sound Listening Group 2 — This group consisted of 15 infants with 33-36,6 GW. A total of one hour of noise measurement was made inside and outside the incubator before, during and after the procedure. The babies were listened to the sound obtained in 3 time periods. If the baby is fed enterally, the feeding of the baby was completed at 10.15/13.00/16.15 before the application, the baby was placed in the prone position and the baby was rested for 30 minutes to ensure gastric emptying. Before the procedure, the baby was watched with a monitor device and recorded on video between 10.45-11.00/13.30-13.45/16.45-17.00. During the baby procedure, uterine sound was listened to the baby in the prone position monitored with a monitor device and recorded on video between 11:00-11.30/13.45-14.15/17.00-17.30 hours. After the procedure, the baby was watched with a monitor device and recorded on video between 11.30-11.45/14.15 and 14.30/17.30-17.45.
  Arms: Intrauterine Sound Listening Group 2

SUMMARY:
Preterm infants lack intrauterine sounds suitable for their development as they are born early. In addition, they are exposed to many unfamiliar sounds for weeks or months in the neonatal intensive care unit (NICU) where their follow-up and care are continued. , one of evidences is that the maternal voices have an effect on the physiological, neurobehavioral and autonomic functions of the preterm infants. Also, the fact that the maternal voice is a non-pharmacological and non-invasive application has importance for the preterm infant. Therefore, considering the optimal well-being of the infant, it is predicted that using the applications that simulate the extrauterine environment of the preterm infant to the intrauterine environment would decrease the stress behaviors of the infants and would provide the physiological values to be followed up in the positive direction, and as a result of these, it would contribute to supporting the recovery and shortening the discharge period. The study was planned as a randomized controlled experimental design in order to determine the effect of the sound applied on the 26-37 week-old preterm infants on their heart rate, oxygen saturation and comfort level.

DETAILED DESCRIPTION:
Preterm infants lack intrauterine sounds suitable for their development as they are born early. In addition, they are exposed to many unfamiliar sounds for weeks or months in the neonatal intensive care unit (NICU) where their follow-up and care are continued. It is known that the preterm infants hear the sounds from the extrauterine and respond to these sounds after the 26th gestational week. The types of the sounds and the level of the noise in the NICU is quite different from the uterus environment. The ambient noise composed of the ventilators, monitors, pagers and alarms of NICU take place of the low-frequency maternal voices in the amniotic environment. For this reason, the preterm infants lack the normal audial stimulants and they are disturbed by the sounds in the NICU environment. As a result, the development of the auditory and language skills and the socio-emotional development of the infants may get harmed. The recent evidences have suggested that the auditory learning and voice recognition experiences of the infants are based on their prenatal experiences. Therefore, it is quite important to make the preterm infants listen to their mothers' voice and the heart rate sound which they are lack of due to their preterm birth and therefore keeping them away from the sounds of the NICU environment.

In the light of this information, one of evidences is that the maternal voices have an effect on the physiological, neurobehavioral and autonomic functions of the preterm infants. Also, the fact that the maternal voice is a non-pharmacological and non-invasive application has importance for the preterm infant. Therefore, considering the optimal well-being of the infant, it is predicted that using the applications that simulate the extrauterine environment of the preterm infant to the intrauterine environment would decrease the stress behaviors of the infants and would provide the physiological values to be followed up in the positive direction, and as a result of these, it would contribute to supporting the recovery and shortening the discharge period.

ELIGIBILITY:
Inclusion criteria:

* Being at -26-36,6 GW,
* In the first week after birth,
* Absence of a congenital anomaly,
* Not being sedated,
* If the baby has been given eye drops, 4-6 hours have passed,
* 20-30 minutes have passed since the last painful attempt

Exclusion criteria:

* Below 26 GW or above 37 GW,
* Absence in the first week after birth,
* Having a congenital anomaly,
* Being sedated,
* The baby is receiving phototherapy

Ages: 26 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Newborn Comfort Behavior Scale (COMFORTneo) | 5 minutes
  The comfort scale (CS) is a scale developed by Ambuel et al., (1992) in order to assess the distress of the children taking the mechanic ventilation support and followed up in the pediatric intensive care unit. The scale was revised by Van Dijk et al. (2009) and developed only for assessing behaviors in the newborns without the physiological parameters. While the lowest score to be obtained from the scale is 6, the highest score is 30. A high score indicates that the infant does not feel comfortable and needs interventions to provide comfort and also 4-6 points indicate moderate pain and distress and 7-10 points indicate severe pain and distress. Kahraman et al., (2014) conducted the Turkish validity and reliability study of the scale with the infants of 24-42 GW.
Heart rate | 1 minutes
  The heart rate of the infants will measured as monitorized.
Peripheral oxygen saturation level | 1 minutes
  The peripheral oxygen saturation level of the infants will measured as monitorized.
Noise level | 1 minutes
  Noise measurement will be made with noise meter from the outside of the incubator during the hours when the study would be conducted.
Sound level | 1 minutes
  In order for the baby to hear the sound created in the incubator; Before each procedure, a noise measuring device was placed in the incubator and the level of sound heard by the baby in the incubator was recorded as dBA. Then the Mp3 device is set to the appropriate volume.

CONTACTS AND LOCATIONS:
Overall Officials: Müjde ÇALIKUŞU İNCEKAR, PhD, Principal Investigator — Yuksek Ihtisas University; Gökhan DENEÇ, PhD, Principal Investigator — Istanbul Technical University; Ayhan TAŞTEKİN, MD, Principal Investigator — Medipol University
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)